CLINICAL TRIAL: NCT03199248
Title: A New Surgical Treatment Technique "Aspiration and Percutaneous Capsulotomy" for Digital Mucous Cyst
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-05-012AC
Record Dates: First submitted 2017-05-30; First posted 2017-06-26 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Digital Mucous Cyst
Keywords: Digital Mucous Cyst; capsulotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the participant accepted needle assisted capsulotomy for DMC
  Interventions: Procedure: Aspiration with percutaneous capsulotomy For digital mucous cysts
- the participant accepted aspiration for DMC only
  Interventions: Procedure: Aspiration with percutaneous capsulotomy For digital mucous cysts

INTERVENTIONS:
Procedure: Aspiration with percutaneous capsulotomy For digital mucous cysts — The surgical procedure for DMCs was using a 18G needle performing aspiration first and then cutting the stalk tract by the needle tip for capsulotomy. All procedure were done with anesthesia. After operation, we asking patient using dressing to pressure the wound about 10 mins to stop bleeding. Later on, the wound was covering with antimicrobial oint(Neomycin) and simple dressing. Educating patient from water for 24 hr.
  Other Names: Aspiration without percutaneous capsulotomy For digital mucous cysts

SUMMARY:
Digital mucous cysts (DMCs) are a benign rubbery cystic lesion which usually involve the dorsal or lateral side of DIP joint (digital interphalangeal joint) or proximal nail fold. The most successful treatment way is surgical management. However, which may cost time, require expertise, may cause infection, prolong wound healing and sometimes may lead to the joint movement limitation. The investigator bring this new technique: percutaneous capsulotomy for digital mucous cysts, which is easy and quick, last but not least, low recurrence rate.

DETAILED DESCRIPTION:
Participant

Between 2016 and 2017, 50 participants with DMCs in Taipei veteran general hospital were included in this study. According to the clinical assessment at OPD(out participants department), DMC was diagnosed. Serial related serial clinical features of DMCs were investigated including participant's age, location, size of cysts, symptoms, duration, nail bed condition, underlying disease(ex. rheumatoid disease, Diabetes) and previous treatment. After explaining to participants about the treatment choice (surgical excision, aspiration of cystic contents, and our needle assisted percutaneous capsulotomy for mucous cyst) and participants agreed with accepting needle assisted percutaneous capsulotomy, they were selected for accepting our needle assisted percutaneous capsulotomy for mucous cyst.

Surgical capsulotomy procedure.

The surgical procedure for DMCs was using a 18G needle performing aspiration first and then cutting the stalk tract by the needle tip for capsulotomy. All procedure were done with local anesthesia. After operation, the investigator asking participants using dressing to pressure the wound about 10 minutes to stop bleeding. Later on, the wound was covering with antimicrobial ointment (neomycin) and simple dressing. Educating participants from water for 24 hrs.

Clinical assessments

The investigator evaluating participant's prognosis by VAS, the improvement of fingernail deformity, the participants' subjective satisfaction and the recurrences was evaluating during follow-ups. This clinical study's approval was obtained from Association of IRB, Taipei veteran general hospital.

ELIGIBILITY:
Inclusion Criteria:

* According to the clinical assessment at OPD(out patient department), DMC was diagnosed. Serial related serial clinical features of DMCs were investigated including pateint's age, location, size of cysts, symptoms, duration, nail bed condition, underlying disease(ex. rheumatoid disease, Diabetes) and previous treatment

Exclusion Criteria:

* autoimmune disease related diffused arthritis, age younger than 20 year-old, severe painful deformity of the involved joint.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the clinical assessment at OPD(out patient department), DMC was diagnosed. Serial related serial clinical features of DMCs were investigated including pateint's age, location, size of cysts, symptoms, duration, nail bed condition, underlying disease(ex. rheumatoid disease, Diabetes) and previous treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
the lesion recurrent or not | 6 months(first evaluation)
  6 months later, DMCs recurrence or not.

SECONDARY OUTCOMES:
Questionnaire | 3 month after treatment(first evaluation)
  The questionnaire including: satisfaction, joint stiffness, nail deformity, pain score(VAS), pigmentation of the lesion site.
Questionnaire | 6 month after treatment(second evaluation)
  The questionnaire including: satisfaction, joint stiffness, nail deformity, pain score(VAS), pigmentation of the lesion site.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei veteran general hospital, Taipei, Taiwan